CLINICAL TRIAL: NCT02035748
Title: Assessment of Anatomical and Functional Outcomes in Patients Treated With Ocriplasmin for Vitreomacular Traction/Symptomatic Vitreomacular Adhesion (VMT/sVMA)
Brief Title: Assessment of Patients Treated With JETREA® for Vitreomacular Traction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-13-056; 2013-005464-25 (EudraCT Number)
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Vitreomacular Traction; Vitreomacular Adhesion
Keywords: Vitreomacular traction; Symptomatic vitreomacular adhesion; Ocriplasmin; JETREA
MeSH Terms: interventions — microplasmin; Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ocriplasmin (Experimental): Ocriplasmin 0.125 mg in a 0.1 mL volume administered as a single dose by intravitreal injection
  Interventions: Drug: Ocriplasmin

INTERVENTIONS:
Drug: Ocriplasmin — 0.5 mg/0.2 mL solution for injection
  Other Names: JETREA®

SUMMARY:
The purpose of this study is to observe the anatomical and functional outcomes of ocriplasmin (JETREA®) over a 6-month follow-up period.

DETAILED DESCRIPTION:
After receiving a single intravitreal injection as per country's product label (Day 0), subjects were followed for a 6-month period (Day 180).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vitreomacular traction/symptomatic vitreomacular adhesion (VMT/sVMA), with evidence of focal VMA visible on Spectral Domain Optical Coherence Tomography (SD-OCT).
* Read, sign, and date an Institutional Review Board/Ethics Committee-approved informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Hypersensitivity to ocriplasmin or any of the JETREA® excipients.
* Active or suspected intraocular or periocular infection.
* Presence of Epiretinal Membrane (ERM) over the macula at baseline.
* Broad VMT/VMA >1500 microns at baseline.
* History of vitrectomy in the study eye.
* History of laser photocoagulation to the macula in the study eye.
* Any relevant concomitant ocular condition that, in the opinion of the investigator, could be expected to worsen or require surgical intervention during the study period.
* Macular hole of >400µm diameter in the study eye.
* High myopia in the study eye.
* Pseudo-exfoliation, Marfan's syndrome, phacodonesis or any other finding in the Investigator's opinion suggesting lens/zonular instability.
* Aphakia.
* History of retinal detachment.
* Diabetic retinopathy, ischaemic retinopathies, retinal vein occlusions.
* Recent ocular surgery or ocular injection.
* Vitreous hemorrhage.
* Exudative age-related macular degeneration (AMD).
* Therapy with another investigational agent within 30 days prior to Visit 1.
* Active, simultaneous enrollment in another ophthalmology clinical study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr Clinical Manager, Ophtha-GCRA, Study Director — Alcon, a Novartis Company

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 87 study centers located in Europe and Canada (10 Italy, 5 Netherlands, 4 Poland, 4 Portugal, 12 Spain, 15 United Kingdom, 3 Belgium, 12 France, 9 Germany, 5 Hungary, and 8 Canada).
Pre-assignment Details: Of the 628 enrolled, 160 subjects were exited prior to initiation of treatment. This reporting group includes all treated subjects (468).
Period: Overall Study
Arm/Group | Ocriplasmin
Started | 468
Completed | 448
Not Completed | 20
Not completed — Adverse Event | 5
Not completed — Death | 3
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 6
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were exposed to the Investigational Product (IP) (Safety Analysis Set).
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345
  Male | 123

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Nonsurgical Resolution of Focal Vitreomacular Traction (VMT/VMA) at Day 28, as Determined by Central Reading Center (CRC) Spectral Domain Optical Coherence Tomography (SD-OCT) Evaluation
Description: Vitreous separation was assessed by SD-OCT using scores ranging from 1 (vitreous attached from macula to ON; separated elsewhere cannot determine foveal) to 12 (unable to determine state of separation). Nonsurgical resolution was defined as a change from baseline score of 5/6/8 to 7/9/10 at Day 28. The assessment of resolution of VMT/sVMA was based upon the anatomical resolution of VMA only, i.e. no resolution of the related symptoms was considered. Thus, the term VMA is used interchangeably with VMT/sVMA. Proportion of subjects is presented as a percentage, with percentage based on the number of subjects who have VMT/sVMA at baseline and SD-OCT value at Day 28. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 28
Population: This analysis population includes all subjects who received treatment with IP and had at least one post-treatment measurement of SD-OCT (FAS). Missing data imputed using the last observation carried forward (LOCF) method. Subjects who had vitrectomy after VMT/sVMA resolution were considered as 'no resolution' after timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 466
percentage of subjects | 47.4

2. Secondary Outcome: Nonsurgical Change From Baseline in Best-corrected Visual Acuity (BCVA) at Distance
Description: BCVA (with spectacles or other visual corrective devices) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) testing at 4 meters. The charts contain 14 rows of letters. BCVA was calculated as the number of letters read correctly and improvement defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 28, Day 90, Day 180
Population: Full Analysis Set. Missing data imputed using LOCF. BCVA values after a vitrectomy were imputed with the last non-missing value prior to the vitrectomy.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 448
letters
  Change from baseline at Day 28 | 1.7 (6.70)
  Change from baseline at Day 90 | 3.0 (7.07)
  Change from baseline at Day 180 | 3.5 (7.77)

3. Secondary Outcome: Proportion of Subjects With Nonsurgical Closure of Macular Hole (MH), if Present at Baseline
Description: The closure of macular hole (a full thickness defect of the retinal tissue involving the anatomical fovea) is defined as a flattened and reattached hole rim along the whole circumference of macular hole. Closure was determined by SD-OCT evaluation and the percentage of subjects tabulated. Proportion of subjects is presented as a percentage, with percentage based on the number of subjects who had macular hole at baseline and OCT value at each specific visit. One eye (study eye) contributed to the analysis.
Time Frame: Day 28, Day 90, Day 180
Population: Full Analysis Set. Missing data imputed using LOCF. Subjects who had vitrectomy after MH closure were considered as 'no MH closure' after the timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 86
percentage of subjects
  Day 28 | 39.5
  Day 90 | 40.7
  Day 180 | 41.9

4. Secondary Outcome: Proportion of Subjects With Nonsurgical Resolution of VMT/sVMA
Description: Vitreous separation was assessed by SD-OCT using scores ranging from 1 (vitreous attached from macula to ON; separated elsewhere cannot determine foveal) to 12 (unable to determine state of separation). Nonsurgical resolution was defined as a change from baseline score of 5/6/8 to 7/9/10 at Day 90 and Day 180. The assessment of resolution of VMT/sVMA was based upon the anatomical resolution of VMA only, i.e. no resolution of the related symptoms was considered. Thus, the term VMA is used interchangeably with VMT/sVMA. Proportion of subjects is presented as a percentage, with percentage based on the number of subjects who have VMT/sVMA at baseline and SD-OCT value at Day 90/Day 180. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 90, Day 180
Population: Full Analysis Set. Missing data imputed using LOCF. Subjects who had vitrectomy after VMT/sVMA resolution were considered as 'no resolution' after the timepoint of vitrectomy.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 466
percentage of subjects
  Day 90 | 47.9
  Day 180 | 49.4

5. Secondary Outcome: Proportion of Subjects Experiencing Pars Plana Vitrectomy (PPV) at Day 180
Description: Pars plana vitrectomy (the surgical removal of vitreous gel from the eye) was captured in Concomitant Ocular Procedures. Proportion of subjects is reported as a percentage. One eye (study eye) contributed to the analysis.
Time Frame: Day 180
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 466
percentage of subjects | 12.0

6. Secondary Outcome: Mean Nonsurgical Change From Baseline in Central Foveal Thickness (CFT)
Description: Nonsurgical change in central foveal thickness (CFT values after a vitrectomy were imputed with the last non-missing value prior to the vitrectomy) was determined by subtracting the measurements in subretinal fluid and retinal pigment epithelium (RPE) elevations and/or SHRM (subretinal hyper-reflective material, such as choroidal neovascularization (CNV)) from the value in total retinal measurement. A lower CFT indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 28, Day 180
Population: Full Analysis Set. Missing data is imputed using LOCF. CFT values after a vitrectomy were imputed with the last non-missing value prior to the vitrectomy.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Ocriplasmin
Number analyzed (Participants) | 466
micrometers
  Baseline (Day 0), n=466 | 276.1 (166.4)
  Change from baseline at Day 28, n=465 | -43.2 (113.47)
  Change from baseline at Day 180, n=466 | -45.4 (131.84)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 7 months). Ocular AEs are presented for both study eye and non-study eye combined. AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject regardless of the causal relationship to the study medication. AEs could be volunteered or solicited by the Investigator or study personnel.
Groups:
- Pretreatment: All subjects consented to participate in the study prior to the initiation of study treatment
- Ocriplasmin: All subjects exposed to the investigational product
Arm/Group | Pretreatment | Ocriplasmin
Serious Adverse Events (participants affected / at risk) | 1/628 | 46/468
Other Adverse Events (participants affected / at risk) | 1/628 | 247/468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=628) | Ocriplasmin (N=468)
Eye operation (Surgical and medical procedures) | 1 | 0
Macular Hole (Eye disorders) | 0 | 8
Hip arthroplasty (Surgical and medical procedures) | 0 | 2
Cardioversion (Surgical and medical procedures) | 0 | 1
Ear operation (Surgical and medical procedures) | 0 | 1
Heart valve replacement (Surgical and medical procedures) | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 1
Lithotripsy (Surgical and medical procedures) | 0 | 1
Renal stone removal (Surgical and medical procedures) | 0 | 1
Shoulder operation (Surgical and medical procedures) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Colonoscopy (Investigations) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 5
Retinal detachment (Eye disorders) | 0 | 4
Vitreous adhesions (Eye disorders) | 0 | 2
Ciliary zonular dehiscence (Eye disorders) | 0 | 1
Vitrectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=628) | Ocriplasmin (N=468)
Visual acuity reduced (Eye disorders) | 1 | 127
Photopsia (Eye disorders) | 0 | 104
Vitreous floaters (Eye disorders) | 0 | 78
Vision blurred (Eye disorders) | 0 | 54
Macular oedema (Eye disorders) | 0 | 52
Eye pain (Eye disorders) | 0 | 40
Colour blindness acquired (Eye disorders) | 0 | 26
Photophobia (Eye disorders) | 0 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.